CLINICAL TRIAL: NCT03329482
Title: Effect of Pulse Ultrasound and Kneading Massage Using Lofnac -Gel in the Management of NSCLBP
Brief Title: Pulse Ultrasound and Kneading Massage in Non- Specific Chronic Low Back Pain
Acronym: NSCLBP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Obafemi Awolowo University (Other)
Responsible Party: Principal Investigator, Adesola Ojo Ojoawo, Principal Investigator, Obafemi Awolowo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ObafemiAU
Record Dates: First submitted 2017-10-30; First posted 2017-11-06 (Actual); Last update posted 2017-11-07 (Actual); Status verified 2017-11

CONDITIONS: Non Specific Low Back Pain
Keywords: Ultrasound; kneading-massage; low back pain; pain intensity; disability
MeSH Terms: conditions — Low Back Pain; Pain | interventions — High-Energy Shock Waves; Massage

STUDY DESIGN:
Intervention Model Description: A total number of 50 subjects were enrolled for the study: 25 subjects for the PUS group and 25 subjects for the KM group in order to give room for attrition. For the purpose of the study the following instruments were used: verbal-rating scale, Roland-Morris disability questionnaire, and an ultrasound machine
Who Masked: Outcomes Assessor
Masking Description: One of the Physiotherapist who carried out the assessment especially when the intervention started did not aware of the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pulse Ultrasound Group A (Experimental): This is the Pulse Ultrasound group. Twenty five patients will be in this group.
  Interventions: Other: PULSE ULTRASOUND
- Kneading Massage Group B (Experimental): This is kneading massage group . Also 25 patients will be in this group.
  Interventions: Other: KNEADING MASSAGE

INTERVENTIONS:
Other: PULSE ULTRASOUND — For group A, The PUS group received pulse mode of ultrasound (sonoplus 490s), with frequency of 1MHZ and intensity of 1.5w/cm according to Ebadi et al 10). Grey's formula was used to estimate the duration of ultrasound (US) for each patient 21). The average local exposure time was one minute and the effective radiating area of the transducer head was 5 cm2. For a patient with an area of low back pain of 40 cm2, the required total treatment time was: 1 min × (40 cm2/5 cm2) = 8 minutes. US was applied using slow circular movements, with the transducer head placed over the painful paravertebral low back region and Lofnac gel used as coupling medium.
  Other Names: ULTRASOUND
  Arms: Pulse Ultrasound Group A
Other: KNEADING MASSAGE — Kneading massage was done with the two hands maintaining a slow circular compression of soft tissues against underlying bone. Pressure was applied as the hands moved proximally, continuously maintaining a contact with the skin, according to Goat22). Lofnac gel was used as a coupling medium for the massage. This was done for an approximately ten and 12 minutes.
  Other Names: MASSAGE
  Arms: Kneading Massage Group B

SUMMARY:
Back pain is one of humanity most frequent complains. About nine of ten adults experience back pain at some points in their life and five out of ten working adults have back pain every year. When continued for long period it may constitute a disability which tries the patient of the most stoical individual as well as the doctor called to bring relief to the suffering victim.

Kneading massage with topical analgesic is a common practice by physiotherapist especially in Nigeria in the management of low back pain, work has been done to know the efficacy of lofnac gel (topical analgesic) via phonophoresis in the management of low back pain(ojoawo,2015), but the comparison of the efficacy of kneading massage and phonophoresis in the management of low back pain has not been well documented. The purpose of this study therefore, is to compare the efficacy of kneading massage and phonophoresis using lofnac gel in the treatment of non-specific chronic low back pain.

DETAILED DESCRIPTION:
The subjects for the study were patients with chronic non-specific low back pain (CNSLBP) receiving treatment at Physiotherapy Department, Osun State Specialist Hospital, Oshogbo, Nigeria. The inclusion criteria for the patients were patients with non-specific low back pain with symptom of pain lasting more than three months. Patients with nerve roots symptoms, underlying systemic or visceral disease, and specific conditions such as neoplasms, fracture, ankylosing spondylitis, previous low back surgery, and pregnancy were excluded from the study. The design of the study was quasi-experimental design.

Among other screening procedures, spinal movements that provoked pain were noted because spinal pain of mechanical origin may be reproduced by movement which induces tension and neural sliding 15). Straight leg raising and Ely's test were carried out according to Nwuga 16) and were found to elicit pain at the lower back. X- ray report of each patient was also reviewed and none of the reports indicated osteoporosis, carcinoma, or pot disease.

In order to determine the number of subjects to be involved, a sample size equation to compare two means according to Eng,17) was used:

N= 4δ2(Zcrit + Zpower)2/D2 Where N is the sample size (the sum of sizes of both comparison group). Where δ is the standard deviation of each group (assumed to have a value of six and to be equal for both groups). Zcrit is the standard normal deviation corresponding to the selective significant criterion [i.e. 0.05 (95% =1.960)].

4 Zpower is the standard deviation corresponding to the selective statistical power (i.e 0.80=0.842).

D is the minimum expected difference between the two mean values, to be significant the value should be 2, therefore D = 5 is chosen .

N=4*62(1.96 + 0.842)2/52 =45.22= 45 Therefore, the total number of 50 subjects were enrolled for the study: 25 subjects for the PUS group and 25 subjects for the KM group in order to give room for attrition. For the purpose of the study the following instruments were used: verbal-rating scale, Roland-Morris disability questionnaire, and an ultrasound machine, among others.

The verbal rating scale (VRS) is a 10-point scale with 1 and 10 indicating the extremes used to assess pain. The VRS was validated with the visual analogue scale by Williamson and Hoggart 18) who concluded that VRS provides a useful alternative to the visual analogue scale scores in the assessment of chronic pain. VRS was used to measure present pain, i.e., pain at the time of study.

Roland Morris Disability Questionnaire (RMDQ): This is a commonly utilised instrument for measuring spinal disability as an outcome measure 19). It is a 24-item questionnaire that is relevant to low back pain disability. RMDQ is easy to score by totalling the sum of circled items (maximum is 24) which represent the final score. The Roland Morris study was referred to as the best single study of assessing short-term outcome of primary care patients with low back pain20).

Ultrasound machine (with pulse and continuous mode; Sonopuls 490, Enraf-Nonius B.V., Rotterdam, The Netherlands): This was used to produce the ultrasonic wave for phonophoresis.

Subjects were randomized into the two groups as follows: Envelopes which contained alphabets A and B were made. Subjects were asked to pick from the envelopes. All subjects who picked A were assigned to ultrasound (PUS) group, whereas subjects who picked B were assigned to kneading massage (KM) group.

Ethical approval was obtained (HREC No: IPHOAU/12/784) from the Health Research and Ethics Committee, Institute of Public Health, Obafemi Awolowo University, Ile-Ife, Nigeria, and informed consent of the participant was obtained.

5 Subjects in each group received 12 sessions of treatment within a period of six weeks of treatments. Subjects in each group were placed on stabilization exercise for 20 minutes. Pulse ultrasound was administered for the subjects in pulse ultrasound group and kneading massage for the control group. Lofnac gel was used as topical gel for the subjects in the two groups. Treatment was administered twice (Monday and Fridays of every week for six weeks). Assessment was done before the treatment began and every Mondays of the week of the treatment.

The PUS group received pulse mode of ultrasound (sonoplus 490s), with frequency of 1MHZ and intensity of 1.5w/cm according to Ebadi et al 10). Grey's formula was used to estimate the duration of ultrasound (US) for each patient 21). The average local exposure time was one minute and the effective radiating area of the transducer head was 5 cm2. For a patient with an area of low back pain of 40 cm2, the required total treatment time was: 1 min × (40 cm2/5 cm2) = 8 minutes. US was applied using slow circular movements, with the transducer head placed over the painful paravertebral low back region and Lofnac gel used as coupling medium.

Kneading massage was done with the two hands maintaining a slow circular compression of soft tissues against underlying bone. Pressure was applied as the hands moved proximally, continuously maintaining a contact with the skin, according to Goat22). Lofnac gel was used as a coupling medium for the massage. This was done for an approximately ten and 12 minutes.

For stabilization exercise, a supervised exercise program was employed for each patient. The exercises included posterior pelvic tilts, sit-ups, bridging, quadruped exercises, and posterior hip and knee muscles stretching 23). Not all patients could do all the exercise at a stretch; exercises were done according to the levels of tolerance and endurance of each patient. Patients were instructed to perform two to three stretches (of all muscles) per treatment and hold the stretch for 20 seconds unless it hurts. Strengthening exercises started with five repetitions and progressed according to each patient's improvement, to three sets of 10 repetitions 10).

In order to avoid co-interaction, subjects were informed not to participate in any other exercise or treatment program until the end of the follow-up period. Also they were informed not to take any analgesic drug during the period of this treatment without the consent of the researchers. However, no patients requested for additional medication apart from the treatment in the department. The primary measure was pain intensity and the secondary outcome measure was disability index. They were measured by a separate physiotherapist who was independent 6 of the study every week of the treatment. Data for pre-treatment, third week, and six week of treatment were used for data analysis.

The data was analyzed using Statistical Package for Social Sciences (SPSS 17). Descriptive statistics and inferential statistics were used to summarize the data. Independent-t-test was used to compare the anthropometric indices of subjects in each group. Repeated measure analysis of variance (ANOVA) was used to compare the mean values of pre-treatment, third-week and sixth-week pain intensity and physical function within the group and across the group. Post hoc analyses were carried out when necessary. An alpha level of <0.05 is set as significant level.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mechanical low back pain who have had pain for more than three months were eligible for the study.

Exclusion Criteria:

* Patients with nerve roots symptoms, underlying systemic or viscera disease and specific condition such as neoplasm, fracture, ankylosing spondylolytis, previous low back surgery and pregnancy were excluded

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-08-12 (Actual); Primary Completion 2017-04-15 (Actual); Study Completion 2017-04-15 (Actual)

PRIMARY OUTCOMES:
The verbal rating scale | 6 Weeks
  The verbal rating scale is a 10-point rating scale that measures present pain intensity of patients. The scale started from 0 and ends with 10. 0 indicate no pain, 1 indicate minimal pain while 5 indicates moderate pain and 10 indicates the most difficult pain called excruciating pain

SECONDARY OUTCOMES:
Roland Morris Disability Questionnaire | 6 weeks
  Roland Morris Disability Questionnaire . It is used to measure disability. It is a 24-item questionnaire that is relevant to low back pain disability. It is scored by totalling the sum of circled items by the patients (maximum is 24) which represent the final score. The score can therefore vary from 0 to 24. 0 indicate no disability and 24 indicates worst disability. The total number of marked statements are added by the clinician. Clinical improvement over time can be graded based on the analysis of serial questionnaire scores. If, for example, at the beginning of treatment, a patient's score was 12 and, at the conclusion of treatment, her score was 2 (10 points of improvement), we would calculate an 83% (10/12 x 100) improvement.

CONTACTS AND LOCATIONS:
Locations (1):
- Obafemi Awolowo University, Ile-Ife, Osun State, Nigeria

IPD SHARING:
Plan to Share IPD: No
The study is planned to be published in a reputable journal. The raw data will be kept in the achieve of theUniversity

REFERENCES:
- [Background] Ebadi S, Ansari NN, Naghdi S, Jalaei S, Sadat M, Bagheri H, Vantulder MW, Henschke N, Fallah E. The effect of continuous ultrasound on chronic non-specific low back pain: a single blind placebo-controlled randomized trial. BMC Musculoskelet Disord. 2012 Oct 2;13:192. doi: 10.1186/1471-2474-13-192. PMID 23031570
- [Background] Goats GC. Massage--the scientific basis of an ancient art: Part 1. The techniques. Br J Sports Med. 1994 Sep;28(3):149-52. doi: 10.1136/bjsm.28.3.149. PMID 8000809
- [Background] Williamson A, Hoggart B. Pain: a review of three commonly used pain rating scales. J Clin Nurs. 2005 Aug;14(7):798-804. doi: 10.1111/j.1365-2702.2005.01121.x. PMID 16000093